CLINICAL TRIAL: NCT04760340
Title: TELUS in Cardiac Surgery Patients. Effect of CPB and Relation to Postoperative Events (PORE).
Brief Title: TELUS in Cardiac Surgery Patients. Effect of CPB and Relation to Postoperative Events (PORE)Events.
Acronym: TELUSPORE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clinique du Millenaire (Other)
Responsible Party: Principal Investigator, Philippe BURTIN, Head of Anesthesiology Department, Clinique du Millenaire
Other Study IDs: Akomé - 01 - 2021
Record Dates: First submitted 2021-01-24; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transesophageal Lung ultrasound (TELUS) was described for the first time in 2016. The clinical significance and benefits for the patient of the results of a TELUS examination has not been investigated to date.

Since all cardiac surgery with CPB cases in adult patients are performed using a TEE probe to monitor cardiac function, a concomitant TELUS examination is possible in all cases.

The study seeks to describe the incidence and severity of the modifications of the aeration of both lungs assessed by TELUS in the perioperative period of adult cardiac surgery and to establish the relation of the TELUS findings with the occurence of postoperative respiratory events (PORE).

Eventually, the study will also provide results about the interobserver variation of the TELUS examination for which there no reference to date.

DETAILED DESCRIPTION:
Trans Esophageal Lung Ultrasound (TELUS) score in Cardiac surgery (CS) patients.

Effect of CPB and relationship between changes on TELUS score and postoperative respiratory events (PORE).

International recommendations for LUS assessment are available as well as the LUS methodology and nomenclature are widely accepted (1). Additionally, transthoracic LUS demonstrated a predictive value for postoperative pulmonary complication in non-cardiac surgery (2).

More recently, the Trans Esophageal Lung Ultrasound (TELUS) has been described (3).

Adult cardiac surgery patients are at special risk of perioperative respiratory complications including pulmonary edema, Acute Respiratory Distress Syndrome (ARDS), prolonged ventilation and non-invasive ventilation (NIV), tracheotomy and pulmonary infection (4). These complications are responsible for a substantial part of the perioperative case fatality rate. Prevention of these complications by using low tidal volume and an open lung strategy has failed to significantly reduce the incidence of postoperative respiratory events (PORE) (5).

A worsening of the TELUS imaging occurs after CPB when compared with pre CPB imaging has been observed. These observations are consistent with the increase of extra vascular lung water during CPB along with specific effects of CPB on lung vessels (6).

Our primary hypothesis is that CPB induced changes in the TELUS imaging score. Our secondary hypothesis is that magnitude of modifications are related to post-operative respiratory events (PORE) and postoperative complications. The TELUS modifications could have a predictive value for post-operative PORE and thus may help to discriminate patients at risk for PORE.

Objectives 1 - Primary objective :

1 - 1 Describing the incidence and severity of the changes in TELUS imaging between the pre CPB and the post CPB assessment.

1. - 2 Describing the relation of the post CPB TELUS findings and the occurrence of PORE during hospital stay. The primary end-point will be a composite of prolonged NIV (> 12 hours) and / or return to Mechanical Ventilation (MV) after a first successful extubation and / or ICU readmission after a first successful ICU discharge. The secondary endpoints will be : total MV duration, total ICU LOS, total hospital LOS, need for tracheotomy, death from all cause.
2. - Secondary objectives

2 - 1 pre / post CPB TELUS imaging will be assessed by a second examiner allowing us to calculate for the first time the pre / post CPB inter-observer variability of TELUS imaging in adult cardiac surgery. Intra observer variability will be assessed as well.

2 - 2 As a standard transthoracic LUS is performed in all CS patients at admission in the ICU post-operatively, the respective relation of the admission LUS and post-CPB TELUS scores with the first PaO2 / fraction of inspired oxygen (FiO2) (P/F) ratio obtained at admission in the ICU.

Methods This is a single center, non-interventional, observational and prospective study.

The study will be registered at Clinical trials.gov. The study will be conducted according to the STROBE guidelines.

All patients will be informed orally during the mandatory pre-anesthesia interview usually performed the day before surgery. A written information document will be given preoperatively to each patient and filed. Patients will be included at the start of the pre-CPB TEE examination.

1. - Anesthesia Briefly, Two standard anesthesia protocols are in use in the institution. Anesthesia will be maintained either with Total Intravenous Anesthesia (TIVA) (continuous infusion of propofol and remifentanil with titration to keep the Bispectral index (BIS) values between 50 and 60) or inhalation anesthesia (remifentanil infusion and continuous sevoflurane inhalation including during CPB). Full muscle relaxation will be obtained with standard doses of atracurium or cisatracurium. Lungs will be ventilated with a low tidal volume of 6 ml.kg-1 (IBW). Standard arterial and central venous catheterization will be inserted in all patients. Hemodynamic monitoring will be performed with a Flotrac sensor and EV1000 monitor (EDWARDS Life Science - Irvine - USA). A continuous airway pressure of 5 cmH2O will be maintained during CPB. After skin closure, patients will be transferred to the ICU and anesthesia infusions will be discontinued after 2 hours if extubation criteria are met : bleeding < 200 ml, normal ECG recording, normal gas exchange, hemodynamic stability with or without low dose vasopressive support (norepinephrine < 100 µg.kg-1.h-1 IV).
2. - CPB CPB will be performed according to institutional standard of care and international guidelines (7) CPB flow will be performed using a centrifugal pump after caval and aortic canulation. In some cases femoral or bicaval canulation will be used. Full anticoagulation will be performed with unfractioned Heparin with POC monitoring (target Activated clotting Time (ACT) : 480 sec) according to guidelines. A minimum of 2.5 l/min CPB flow will be maintained. Cardioplegia will be performed by antegrade and/or retrograde normothermic cardioplegia according to the type of surgery. Centrifugation of the residual volume of the CPB circuit at the end of the procedure will be performed and re-transfused to the patient.
3. - TEE Comprehensive TEE will be performed in anesthetized patients before skin incision (preCPB) and after chest closure (post CPB) using a GE Vivid S7 ultrasound system (GE Healthcare, Chicago IL, USA). TEE examination will be performed according to our standard procedure, reporting and archiving. Pre and post CPB LV function indices (LVEF, E wave, A wave velocities, E' and S'Lat velocities, quantification of Mitral Regurgitation (MR) if present).
4. - TELUS Using the same imaging system, TELUS will be performed pre and post CPB according to the method described by previous authors (3). Sagittal (90°) mid-esophageal view and rotation of the probe will allow right lung interrogation of the anterior (60° rotation), lateral (90° rotation) and posterior (120° rotation) zones and left lung interrogation of the anterior (300° rotation), lateral (270° rotation) and posterior (240° rotation) zones. For each zone a TELUS score will be defined according to standard definitions : TELUS 0 : presence of A lines, TELUS 1 : less than 3 B lines , TELUS 2 : more than 3 B lines or confluent B lines, TELUS 3 : sub pleural condensation. Additionally, immediate findings (Pleural effusion, Alveolar consolidation, Pneumothorax) will be recorded.

   Thus, the maximum LUS score per lung will be 9 and the maximum LUS score per patient will be 18.
5. - LUS A transthoracic LUS examination will be performed immediately after arrival in the ICU (standard routine practice). For each lung the anterior, lateral and posterior zones will be interrogated. For each zone a LUS score will be defined according to standard definitions : LUS 0 : presence of A lines, LUS 1 : less than 3 B lines , LUS 2 : more than 3 B lines or confluent B lines, LUS 3 : sub pleural condensation. Additionally, immediate findings (Pleural effusion, Alveolar consolidation, Pneumothorax) will be recorded.

   Thus the maximum LUS score per lung will be 9 and the maximum LUS score per patient will be 18.
6. - Biological data

   Arterial blood gas are routinely drawn as a standard practice :

   a - After anesthesia and before skin incision b -Immediately after obtaining the CPB full flow c - Every 20 - 25 min during CPB d -5 - 10 min after protamine injection. e - 15 min after arrival in the ICU

   a,d, and e blood gases results will be recorded and P/F ratio will be calculated.

   Troponin will be measured (ROCHE Diagnostics, Basel, Switzerland) in all patients at H24 as an institution standard practice.
7. - Recorded data

   All data will be recorded in an anonymous database (EXCEL worksheet). The recorded data will be:
   * Hospital file number, initials, Demographic and procedural data, comorbidities, medications, baseline hematocrit and creatinine level
   * Pre CPB TELUS data and score, TEE data, P/F, MAP, SAP, DAP, Heart Rate, O2 arterial saturation
   * post CPB TELUS data and score, TEE data, P/F, MAP, SAP, DAP, Heart Rate, O2 arterial saturation, total IV fluid balance during CPB.
   * LUS data and score, P/F after arrival in the ICU
   * Post-operative respiratory events (PORE) : time to extubation (hours), total time on NIV (hours), return to mechanical ventilation (intubation), total time on ventilation (hours),Tracheotomy and duration (hours), length of stay (LOS) in ICU (hours), pneumothorax after removal of chest tubes, pleural effusion, pneumonia (≥ 2 criteria including fever> 38.5 ° C or T <36 ° C, leukocytosis> 109/ L , purulent tracheal secretions and the appearance or persistence of an infiltrate on the CXR), atelectasis, pulmonary embolism, NO inhalation and total duration (hours), ARDS (Berlin definition), sternal wound infection, in-hospital LOS (days)
   * Other in-hospital complications : cardiac ischemia, congestive heart failure, ventricular dysrhythmia, new onset of atrial fibrillation (NOAF), Acute kidney failure (AKI), Renal replacement therapy (RRT) and total duration (hours), cerebral ischemia, sepsis from other origin than the lungs, blood transfusion (units count), ICU Readmission, death from all cause.
8. - Statistical analysis As there is no previous study that have observed TELUS during CPB in CS, sample size calculation cannot be done because mean score and standard deviation are not known. All patients with complete TELUS and LUS examinations during a four month period will be included.

Inter-observer variability will be assessed using the Bland Altman method (8), Lin test (9), and weighted kappa test (10).

Qualitative variables will be expressed as an absolute value and percentage. Quantitative variables will be expressed as a mean and Standard deviation (SD) or median and interquartile range depending on the normality of the data distribution.

Comprehensive descriptive statistics. Comparisons will be made between the pre and post CPB TELUS recordings for demographic, procedural and biological data.

Two groups will be defined according to the value of the PostCPB TELUS Score. Group HITELUS with the patients with TELUS score of 12 or higher. Group LOTELUS with the patients with TELUS score under 12. The two groups will be compared for the incidence of the primary and secondary outcomes and for all comorbidities and procedural variables.

Comparisons will be made between the post CPB TELUS and ICU LUS recordings for demographic, procedural and biological data.

A composite score of PORE will be built. To determine TELUS / LUS variables associated with PORE occurrence, multivariate logistic regression will be performed.

To determine the predictive performance of TELUS / LUS scores for RE occurrence ROC curves will be generated with calculation of Area Under the Curve (AUC) with confidence intervals, Se, Sp, positive and Negative predictive values (PPV and NPV), Youden index values.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgery patients with a comprehensive TEE and TELUS examination pre CPB will be included.

Exclusion Criteria:

* Previous lung surgery
* Previous thoracic radiation therapy for cancer (lung, breast, lymphoma or other)
* Mitral valve surgery using a mini thoracotomy and video assistance
* Use of an ultrafiltration device during CPB
* Mechanical ventilation initiated before arrival in the OR.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult cardiac surgery with CPB and TEE monitoring
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Extubation time (minutes) | 150 days
  Time from ICU admission to first postoperative successful extubation.
Total postoperative NIV time (hours) | 150 days
  Total time on NIV during postoperative hospital stay
Total MV time (hours) | 150 days
  Total time on MV during postoperative hospital stay
Total ICU stay (hours) | 150 days
  Length of stay in the icu during hospital stay

SECONDARY OUTCOMES:
Pre CPB TELUS score (n) | 1 day
  Cumulative score of the TELUS grading for the 3 zones of each lung (Min : 0 ; Max : 18) calculated before CPB
Post CPB TELUS score (n) | 1 day
  Cumulative score of the TELUS grading for the 3 zones of each lung (Min : 0 ; Max : 18) calculated after CPB
Post CPB P/F ratio (mmHg) | 1 day
  Ratio between PaO2 (mmHg) and FiO2 (%)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BURTIN, Principal Investigator — Dr Philippe BURTIN

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Zieleskiewicz L, Papinko M, Lopez A, Baldovini A, Fiocchi D, Meresse Z, Boussuges A, Thomas PA, Berdah S, Creagh-Brown B, Bouhemad B, Futier E, Resseguier N, Antonini F, Duclos G, Leone M. Lung Ultrasound Findings in the Postanesthesia Care Unit Are Associated With Outcome After Major Surgery: A Prospective Observational Study in a High-Risk Cohort. Anesth Analg. 2021 Jan;132(1):172-181. doi: 10.1213/ANE.0000000000004755. PMID 32224722
- [Background] Cavayas YA, Girard M, Desjardins G, Denault AY. Transesophageal lung ultrasonography: a novel technique for investigating hypoxemia. Can J Anaesth. 2016 Nov;63(11):1266-76. doi: 10.1007/s12630-016-0702-2. Epub 2016 Jul 29. PMID 27473720
- [Background] Litwinowicz R, Bartus K, Drwila R, Kapelak B, Konstanty-Kalandyk J, Sobczynski R, Wierzbicki K, Bartus M, Chrapusta A, Timek T, Bartus S, Oles K, Sadowski J. In-hospital mortality in cardiac surgery patients after readmission to the intensive care unit: a single-center experience with 10,992 patients. J Cardiothorac Vasc Anesth. 2015;29(3):570-5. doi: 10.1053/j.jvca.2015.01.029. Epub 2015 Jan 16. PMID 26009285
- [Background] Lagier D, Fischer F, Fornier W, Huynh TM, Cholley B, Guinard B, Heger B, Quintana G, Villacorta J, Gaillat F, Gomert R, Degirmenci S, Colson P, Lalande M, Benkouiten S, Minh TH, Pozzi M, Collart F, Latremouille C, Vidal Melo MF, Velly LJ, Jaber S, Fellahi JL, Baumstarck K, Guidon C; PROVECS Study Group. Effect of open-lung vs conventional perioperative ventilation strategies on postoperative pulmonary complications after on-pump cardiac surgery: the PROVECS randomized clinical trial. Intensive Care Med. 2019 Oct;45(10):1401-1412. doi: 10.1007/s00134-019-05741-8. Epub 2019 Oct 1. PMID 31576435
- [Background] Huffmyer JL, Groves DS. Pulmonary complications of cardiopulmonary bypass. Best Pract Res Clin Anaesthesiol. 2015 Jun;29(2):163-75. doi: 10.1016/j.bpa.2015.04.002. Epub 2015 Apr 23. PMID 26060028
- [Background] Authors/Task Force Members; Kunst G, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Puis L, Wahba A; EACTS/EACTA/EBCP Committee Reviewers; Alston P, Fitzgerald D, Nikolic A, Onorati F, Rasmussen BS, Svenmarker S. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Br J Anaesth. 2019 Dec;123(6):713-757. doi: 10.1016/j.bja.2019.09.012. Epub 2019 Oct 2. No abstract available. PMID 31585674
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Lin LI. A concordance correlation coefficient to evaluate reproducibility. Biometrics. 1989 Mar;45(1):255-68. PMID 2720055
- [Background] Banerjee et al. Beyond kappa : a review of interrater agreement measures. Can. J. Statistics 1999 ; 27 : 3 - 23.